CLINICAL TRIAL: NCT01655641
Title: Role of Tranexamic Acid for Reducing Blood Loss in Patients Undergoing Major Gastro-intestinal Surgery
Brief Title: Study of Tranexamic Acid for Reducing Blood Requirement in Patients Undergoing Major Gastro-intestinal Surgery
Acronym: TMGS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr Bikal Ghimire, Assistant Professor, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: # WS2017115
Record Dates: First submitted 2012-07-23; First posted 2012-08-02 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Hepatocellular Cancer; Colon Cancer
Keywords: Blood transfusion; Bleeding; Major Gastro-intestinal surgery; Tranexamic Acid
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Colonic Neoplasms; Hemorrhage | interventions — Tranexamic Acid; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid arm (Experimental): Along with the standard of care (routine surgical care involved in preventing blood loss during surgery) this arm will receive drug Tranexamic acid
  1gm stat, preoperatively (30 mins) 10mg / kg body weight, 8 hourly for 5 days via IV for non-renal impaired subjects.
  Alternate IV dosing for renally-impaired subjects: 10mg/Kg BID (1.36 - 2.83 mg/dl clearance); 10mg/Kg QD (2.84 - 5.66 mg/dl clearance; and 10mg/Kg Q48H or 5mg/Kg (.5.66mg/dl clearance)
  Interventions: Drug: Tranexamic acid
- Standard of care arm (Active Comparator): Includes routine surgical care involved in preventing blood loss during and after surgery.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Tranexamic acid — Drug: Tranexamic acid
  1gm stat, preoperatively (30 mins) 10mg / kg body weight, 8 hourly for 5 days via IV For non-renal impaired subjects.
  Alternate IV dosing for renally-impaired subjects: 10mg/Kg BID (1.36 - 2.83 mg/dl clearance); 10mg/Kg QD (2.84 - 5.66 mg/dl clearance; and 10mg/Kg Q48H or 5mg/Kg (.5.66mg/dl clearance)
  Other Names: Cyklokapron®
  Arms: Tranexamic acid arm
Other: Standard of care — Includes routine surgical care involved in preventing blood loss during and after surgery.
  Arms: Standard of care arm

SUMMARY:
Primary objective of the study is to compare requirement of blood transfusion and mortality in patients receiving Tranexamic acid (Cyklokapron®) and those not receiving it.

Secondary objective is to; assess the re-bleeding events; need for surgical intervention; length of stay in Intensive care unit in between the two groups.

DETAILED DESCRIPTION:
Background:

Surgery is one of the major causes of blood loss. Though major blood loss is associated with cardiovascular procedures, liver transplantation etc, transfusions are frequently required in major gastrointestinal surgeries such as Whipples Procedure; Liver resections etc.1 Transfusion is associated with numerous risks such as mismatched transfusion, allergic reactions, transmission of infections, and acute lung injury etc.2 Though transfusion can be life saving, it is essential to rationalize transfusion whenever possible.

A number of agents have been tried in the past that stabilizes the coagulation system in the body minimizing blood loss; an ideal agent is yet to be found. Tranexamic acid, {trans-4-(aminomethyl) cyclohexanecarboxylic acid} is a competitive inhibitor of plasminogen activation, and at much higher concentrations, a noncompetitive inhibitor of plasmin.3 Tranexamic acid was first approved by the FDA in 1986 as an injection, under the brand name Cyklokapron®. This agent has been in use for last 40 years in many traumatic conditions with various successes with waxing and waning of its use. There has been a resurgence of interest in its use lately as more is known of this molecule. Tranexamic acid has been found to be very effective in orthopedic surgeries.4,5,6 A Cochrane review on 'antifibrinolytic use for minimizing perioperative blood transfusion' involving 21 trails of tranexamic acid vs. control in patients undergoing orthopedic surgery showed significant reduction in blood transfusion and perioperative blood loss.7 Randomized trial of tranexamic acid done on cardiac surgery patients as early as 1996 had shown significant reduction of red-cell transfusion and other blood products.8 CRASH 2 Trial (Clinical Randomization of an Antifibrinolytic in Significant Haemorrhage) is a large placebo-controlled trial studying the effects of early administration of a short course of tranexamic acid on death, vascular occlusive events and blood transfusion in adult trauma patients with significant hemorrhage. It involved 274 hospitals across 40 countries and started in 2005 and concluded that tranexamic acid could safely reduce the risk of death in bleeding trauma patients.9 Intraoperative use of low dose tranexamic acid has been observed to be safe and effective in reducing the rate of perioperative blood transfusions in patients undergoing radical retropubic prostatectomy.10 It has also been approved by FDA for use in menorrhagia.

Though it is being used in gastrointestinal bleeding and abdominal trauma, it is not routinely used in major gastrointestinal surgeries. In this context, this study is undertaken to evaluate the efficacy of tranexamic acid in major gastrointestinal surgeries.

Investigators hypothesize that addition of Tranexamic acid, an antifibrinolytic agent, to conventional therapy will lead to an improved outcome characterized by lower transfusion requirements.

Detailed Description:

After informed consent is obtained patients will be randomized to receive either Tranexamic acid along with the conventional therapy or conventional therapy only. All patients undergoing major gastrointestinal surgery (involving resection of stomach, pancreas, esophagus, colon, liver) will be included for the surgery and this will be decided by the surgeon prior to the surgery. Randomization will be done prior to surgery by the closed envelope method. Tranexamic acid will be administered in a loading dose of 1 gm intravenously over 10 minutes, 30minutes before surgery followed by 10mg / kg body weight, 8 hourly for 5 days. Post operative blood requirements and the fluids in the drain will be monitored along with the HB/PCV level every day for 7 days or until the drains are removed.

Tranexamic acid is an antifibrinolytic agent that has been shown to be associated with reduced bleeding and transfusion requirement in surgical patients. We would like to randomize patients to receive either Tranexamic acid in addition to conventional therapy or the conventional therapy only and monitor outcome. Intraoperative blood requirements are usually governed by the intraoperative blood loss hence, only post operative blood transfusions will be taken as the 'Post operative blood requirements' for these patients. Post operative complications will be assessed according to the Clavien-Dindo Classification system for surgical complications.11,12,13 Patients will be monitored until discharge and after 30 days to assess for any complication. Duration of ICU stay, duration of admission and Mortality will be monitored for both groups of patients.

Requirement for Transfusion will be assessed by the operating surgeon. Patients will be monitored post operatively with the hemoglobin and PCV level and the drain fluid amount and nature. Transfusion will be given for ongoing blood loss at the discretion of the operating surgeon or when hemoglobin level is <8milligram per deciliter hemoglobin or hematocrit value of less than 24 percent in healthy individual or < 10mg/dl in high risk patients.14 Transfusion of Fresh Frozen Plasma (FFP) and Platelet Rich Plasma (PRP) will be done as required.

This study should provide us with information about the efficacy of this medicine in patients undergoing major GI surgery. Data from this trial will provide us information about utility of pursuing this modality of therapy.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing major GI surgery that includes resection of:

* Esophagus
* Stomach
* Spleen
* Liver
* Pancreas
* Colon

Exclusion Criteria:

* Pre op HB less than 10mg/dl
* Pregnant or lactating women
* On anticoagulation therapy
* Patients with history of thromboembolism
* Patients with history of myocardial infarction or ischemic cerebrovascular accident
* Patient with end stage renal disease
* Patients with DNR status
* Patients with known bleeding abnormalities
* Emergency/unplanned surgeries
* Patients with known allergy/contraindications to Tranexamic acid
* Patients not capable of giving consent for medical reasons (psychiatric etc)\
* Patients not giving consent or opting to withdraw from the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Primary objective of the study is to compare transfusion requirements and Mortality in patients receiving Tranexamic acid (Cyklokapron®) and those not receiving it. | 30 days

SECONDARY OUTCOMES:
Secondary outcome measure | 30days
  Re-bleeding events
Secondary Outcome measure | 30 days
  Need for surgical intervention
Secondary outcome measure | 30 days
  Length of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Bikal Ghimire, MS, Principal Investigator — Tribhuvan University, Nepal
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Kathmandy, Nepal

REFERENCES:
- [Result] Mannucci PM, Levi M. Prevention and treatment of major blood loss. N Engl J Med. 2007 May 31;356(22):2301-11. doi: 10.1056/NEJMra067742. No abstract available. PMID 17538089
- [Result] Blajchman MA, Vamvakas EC. The continuing risk of transfusion-transmitted infections. N Engl J Med. 2006 Sep 28;355(13):1303-5. doi: 10.1056/NEJMp068178. No abstract available. PMID 17005947
- [Result] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Result] Colomina MJ, Bago J, Fuentes I. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine 2008; 33: 2577-80. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1740-1; author reply 141. doi: 10.1097/BRS.0b013e3181a9ce1f. No abstract available. PMID 19770617
- [Result] Elwatidy S, Jamjoom Z, Elgamal E, Zakaria A, Turkistani A, El-Dawlatly A. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2577-80. doi: 10.1097/BRS.0b013e318188b9c5. PMID 19011538
- [Result] Urban MK, Beckman J, Gordon M, Urquhart B, Boachie-Adjei O. The efficacy of antifibrinolytics in the reduction of blood loss during complex adult reconstructive spine surgery. Spine (Phila Pa 1976). 2001 May 15;26(10):1152-6. doi: 10.1097/00007632-200105150-00012. PMID 11413430
- [Result] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, McClelland B, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001886. doi: 10.1002/14651858.CD001886.pub2. PMID 17943760
- [Result] Katsaros D, Petricevic M, Snow NJ, Woodhall DD, Van Bergen R. Tranexamic acid reduces postbypass blood use: a double-blinded, prospective, randomized study of 210 patients. Ann Thorac Surg. 1996 Apr;61(4):1131-5. doi: 10.1016/0003-4975(96)00022-7. PMID 8607670
- [Result] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Result] Crescenti A, Borghi G, Bignami E, Bertarelli G, Landoni G, Casiraghi GM, Briganti A, Montorsi F, Rigatti P, Zangrillo A. Intraoperative use of tranexamic acid to reduce transfusion rate in patients undergoing radical retropubic prostatectomy: double blind, randomised, placebo controlled trial. BMJ. 2011 Oct 19;343:d5701. doi: 10.1136/bmj.d5701. PMID 22012809
- [Result] Clavien PA, Sanabria JR, Strasberg SM. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Surgery. 1992 May;111(5):518-26. PMID 1598671
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Practice guidelines for perioperative blood transfusion and adjuvant therapies: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Anesthesiology. 2006 Jul;105(1):198-208. doi: 10.1097/00000542-200607000-00030. No abstract available. PMID 16810012